CLINICAL TRIAL: NCT03467191
Title: Predicting Alcohol Use and Alcohol Use Disorder Symptoms From Subjective Responses to Alcohol in a Laboratory Social Setting
Brief Title: Behavioral Alcohol Responses (BAR) Study
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); University of Pittsburgh (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Kasey Creswell, Associate Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY2017_00000346; R01AA025936 (NIH)
Record Dates: First submitted 2018-03-01; First posted 2018-03-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Drinking; Alcohol Use Disorder; Alcohol Intoxication; Alcohol; Harmful Use; Alcoholism; Binge Drinking
MeSH Terms: conditions — Alcohol Drinking; Alcoholism; Alcoholic Intoxication; Binge Drinking | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol Beverage (Experimental): Moderate dose of alcohol (target BAC .08%)
  Interventions: Drug: Alcohol
- Placebo Beverage (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alcohol — target BAC .08%
  Arms: Alcohol Beverage
Other: Placebo — placebo beverage
  Arms: Placebo Beverage

SUMMARY:
This study aims to identify risk factors that prospectively predict alcohol problems in young adults.

DETAILED DESCRIPTION:
The vast majority of alcohol use takes place in social settings, yet nearly all human experimental work has administered alcohol to individuals in isolation. This study will examine the effects of alcohol in social groups and test whether these responses predict the escalation of alcohol use and development of alcohol use disorder symptoms. Participants will also complete smartphone surveys querying subjective responses to alcohol in their daily lives.

N=400 male and female young adults will participate in a laboratory session with two other participants and will consume either a moderate dose of alcohol or placebo beverage. Subjective and objective responses to alcohol will be assessed. Participants will also complete surveys on their smartphones; these will occur during drinking episodes and at random times throughout the day. Follow-up sessions will occur at 6-months and 12-months, to collect information about drinking habits and potential alcohol-related problems.

ELIGIBILITY:
Inclusion Criteria:

* 21 to 29 years of age
* currently drinks alcohol
* owns a smartphone

Exclusion Criteria:

[Exclusion criteria are masked from public viewing until data collection is complete. Please contact project managers.]

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — May be either male or female, but must be same as gender assigned at birth.
Enrollment: 782 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Alcohol Use at 12-months | 12-month follow-up
  Timeline Follow Back Method
Change from Baseline Alcohol Use Disorder Symptoms at 12-months | 12-month follow-up
  Structured Clinical Interview for DSM-5

SECONDARY OUTCOMES:
Subjective Responses to Alcohol | 1 day (laboratory session) and 21-day ambulatory assessment period
  Participants will indicate how they feel after drinking alcohol using the Brief-Biphasic Alcohol Effects Scale, which is a 6-item scale assessing alcohol's acute stimulant and sedative effects (0-10 scale, with higher scores indicating higher values).
Social Bonding | 1 day (laboratory session)
  Facial expressions of emotions using Paul Ekman's Facial Action Coding System (FACS). The duration of AUs associated with positive and negative affect will be coded.
Social Bonding | 1 day (laboratory session)
  Perceived Group Reinforcement Scale, which is a 12-item scale assessing self-reported bonding (1-9 scale, with higher scores indicating more bonding).
Mood | 1 day (laboratory session)
  8-item Mood Measure, which is an 8-item scale assessing mood items from each of the four quadrants of the affective circumplex (with higher scores indicating more felt emotion).
Alcohol Use | 21-day ambulatory assessment period
  Quantity of standard drinks consumed.

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No